CLINICAL TRIAL: NCT03318926
Title: Increased Amount and Time of Tea Consumption is Associated With a Decreased Risk of Renal Stone Disease in a Taiwanese Population
Brief Title: Increased Tea Consumption is Associated With a Decreased Risk of Renal Stone Disease in a Taiwanese Population
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-ER-106-066
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Renal Stone
Keywords: tea, cup-year, renal stone disease
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The objective of the this study was to examine the amount and duration of tea consumption in relation to the risk of renal stone disease.

DETAILED DESCRIPTION:
Previous studies have investigated the association between tea consumption and renal stone disease, but the results are still unclear. Besides, the impact of the duration of tea consumption has not yet been investigated in the aforementioned studies. The present study was conducted as a retrospective research to investigate the relationship between both tea consumption amount and time and renal stone disease. Information on tea consumption was obtained by four closed-ended questions in questionnaires, and the diagnosis of renal stones was established on the results of abdominal sonography.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old

Exclusion Criteria:

* individuals with a history of hyperuricemia or gout at baseline, findings of abdominal ultrasound showing transplant kidney, only one kidney, or gouty nephropathy, or missing data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: examinees who were ≥ 18 years old and underwent health check-ups with abdominal sonography at the health examination center of National Cheng Kung University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 13842 (Actual)
Dates: Start 2001-06 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Renal stone diseases | health check-ups from June 2001 to August 2009
  The diagnosis of renal stones was established on the results of abdominal sonography